CLINICAL TRIAL: NCT06838637
Title: The Safety and Feasibility of Home-based Non-invasive Spinal Cord Stimulation for Orthostatic Hypotension in Individuals with Severe Autonomic Dysfunctions
Brief Title: Transcutaneous Spinal Cord Stimulation Home Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Berger (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); International Collaboration on Repair Discoveries (Other); SpineX Inc. (Industry); Vancouver Coastal Health (Other Government); University of British Columbia (Other); Rick Hansen Foundation (Other)
Responsible Party: Sponsor-Investigator, Michael Berger, Clinical Assistant Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H23-00192
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Multiple System Atrophy, Parkinson Variant
Keywords: Transcutaneous Spinal Cord Stimulation; SCONE; Orthostatic Hypotension; Bowel Dysfunction; Autonomic Dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Multiple System Atrophy; Hypotension, Orthostatic; Intestinal Diseases; Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcutaneous Spinal Cord Stimulation (Experimental): Transcutaneous spinal cord stimulation (TSCS) will be delivered using a portable non-invasive spinal cord stimulator (SCONE, SpineX Inc., CA, USA).
  Interventions: Device: Spinal COrd NEuromodulation ("SCONE") Device

INTERVENTIONS:
Device: Spinal COrd NEuromodulation ("SCONE") Device — A non-invasive electrical device that provides transcutaneous spinal cord stimulation (TSCS) to the spinal cord by electrodes connected to a battery-powered source.

SUMMARY:
The goal of this pilot clinical trial is to examine the safety and feasibility of SCONE as home based therapy for orthostatic hypotension and bowel dysfunction in individuals with spinal cord injury or multiple system atrophy. The main aims of the study are:

* To establish a safe protocol for home-based transcutaneous spinal cord stimulation therapy at the research centre
* To test the safety and feasibility of home-based transcutaneous spinal cord stimulation therapy on orthostatic hypotension and bowel dysfunction

Participation will last approximately 10 weeks (excluding screening period) and involves

* Attending the study center to collect baseline evaluations and to plan where electrodes will be placed
* A 2 week treatment period at the centre with 3 visits per week
* A 6 week home based therapy period involving 1 hour treatments twice a day
* Attending the study center to collect post-treatment evaluations

DETAILED DESCRIPTION:
Visit 1 - Screening

Visit 2 - Baseline Assessments

Visit 3 - Baseline EMG Mapping of Spinal Cord Segments with transcutaneous spinal cord stimulation

Visits 4-9 - Transcutaneous spinal cord stimulation

HOME-BASED Therapy (6 weeks)

Visit 10 - Post-treatment Autonomic Function Assessments

Visit 11 - Post-treatment Cardiac Function Assessments

ELIGIBILITY:
INCLUSION CRITERIA

* A participant must meet all of the following criteria in order to be eligible for inclusion:

  1. Resident of British Columbia, Canada with active provincial medical services plan
  2. Male or female, 19-70 years of age The safety and feasibility of home-based non-invasive spinal cord stimulation for orthostatic hypotension in individuals with severe autonomic dysfunctions (H23-00192) Protocol Version 1.0, December 8, 2023 Page 6 of 23
  3. Chronic spinal cord injury (SCI) (non-progressive, with complete motor paralysis) at or above the T6 spinal segment OR Multiple System Atrophy (MSA) of the parkinsonian type.
  4. >1-year post injury or diagnosis, at least 6 months from any spinal surgery.
  5. American Spinal Injury Association Impairment Scale (AIS) A, B for SCI or having OH (Orthostatic Hypotension) for MSA.
  6. Willing and able to comply with all clinic visits and study-related procedures.
  7. Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
  8. No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing.
  9. Stable management of spinal cord related clinical issues (i.e., spasticity management).
  10. Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

      10.1. Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit.

      10.2. Women of childbearing potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence.
  11. Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment.
  12. Must provide informed consent.

EXCLUSION CRITERIA

* A participant who meets any of the following criteria will be ineligible to participate:

  1. Ventilator dependent.
  2. Clinically significant, unmanaged, depression (PHQ-9 above 15) or ongoing drug abuse.
  3. Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the participant to participate in this study.
  4. Intrathecal baclofen pump.
  5. Cardiovascular, respiratory, bladder, or renal disease unrelated to spinal cord injury (SCI) or presence of hydronephrosis or presence of obstructive renal stones.
  6. Presence of severe acute medical issue that in the investigator's judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to acute urinary tract infections, active heterotopic ossification, newly changed antidepressant medications [tricyclics], debilitating muscle pain, pressure sores, or unstable diabetes.
  7. Any implanted metal (other than dental implants) in the skull or presence of pacemakers, stimulators, or medication pumps in the trunk.
  8. Takes more than 40mg of Baclofen per day.
  9. Severe anemia (Hgb<8 g/dl or Hgb,80 g/L) or hypovolemia as measured by hematocrit via blood test in the last six months.
  10. Participant is a member of the investigational team or his/her immediate family.
  11. Participant has undergone electrode implantation surgery.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) changes in millimeters of mercury (mmHg) during TSCS | 6 weeks
  Changes in SBP measures will be used to establish the BP component of the safety protocol for home-based TSCS with the purpose to mitigate orthostatic hypotension (OH).
Blood pressure (BP) changes in millimeters of mercury (mmHg) in 24-hrs | 6 weeks
  BP changes will be used to test the safety and feasibility of home-based TSCS (6 weeks) for orthostatic tolerance and bowel function in daily activities. The primary safety and feasibility measures will be continuously measured BP with a wireless BP device (Caretaker Medical LLC, USA, Class II, Medical Device Licence 320275) with and without stimulation, skin condition, any adverse event reports related to the stimulation.

SECONDARY OUTCOMES:
24-hour BP measurement in millimeters of mercury (mmHg) | 6 weeks
  BP data (i.e., systolic BP) will be monitored and used as a secondary safety measure in relation to better understanding OH in the context of the time course of cardiovascular changes in 24-hours.
Cardiovascular monitoring in mmHg | 6 weeks
  Beat-by-beat oscillometric cardiovascular monitoring (i.e., mmHg) will be tracked and used as a secondary safety measure in relation to better understanding OH in the context of the time course of cardiovascular function during the mock home-based sessions.
Adverse events (i.e., abnormal electrocardiograph) | 6 weeks
  Adverse events (i.e., abnormal electrocardiograph) will be tracked and used as a secondary safety measure in relation to better understanding OH in the context of the time course of the frequency and type of adverse events that can occur during mock home-based sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Berger, MD, FRCPC, Principal Investigator — The University of British Columbia; Andrei Krassioukov, MD, FRCPC, Study Director — The University of British Columbia
Locations (1):
- ICORD, Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada